CLINICAL TRIAL: NCT06360835
Title: Our Experience in the Management of Therapeutic Failures of Fractures of the Proximal End of the Femur (About 35 Cases)
Status: Completed | Type: Observational
Sponsor: Ibn Jazzar Hospital (Other)
Responsible Party: Principal Investigator, Zied Mansi, Principal investigator, Ibn Jazzar Hospital
Other Study IDs: IRB00001193
Record Dates: First submitted 2024-03-28; First posted 2024-04-11 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2024-04

CONDITIONS: Proximal Femur Fractures
Keywords: femoral neck fracture; pertrochanteric fracture; internal osteosynthesis; mechanical complications
MeSH Terms: conditions — Proximal Femoral Fractures; Femoral Neck Fractures | interventions — Arthroplasty, Replacement, Hip; Bone Plates

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- cases of recurrent fractures of the proximal end of the femur following surgical treatment failure
  Interventions: Procedure: total hip arthroplasty

INTERVENTIONS:
Procedure: total hip arthroplasty
  Other Names: plate; dynamic condylar screw

SUMMARY:
Osteosyntheses employed in treating fractures at the upper end of the femur play a critical role in facilitating a swift recovery by minimizing immobilization periods and enabling early rehabilitation of the affected joints, thereby promoting a speedy return to normal walking function.

Osteosynthesis alters the mechanical dynamics of the bone segment, which undergoes continual changes during the consolidation and mobilization phases of recovery. Throughout these stages, a range of mechanical complications may arise, posing challenges despite the successful prevention of infections. Non-infectious complications associated with the presence of osteosynthesis materials, especially in weight-bearing areas like the lower limb, remain a concern.

In light of these considerations, surgeons must exercise meticulous care in selecting synthetic materials to mitigate the risk of osteosynthesis failures. In cases where internal fixation fails, the standard recourse often involves converting to total hip arthroplasty (THA).

However, it is essential to note that THA subsequent to complications arising from proximal femur osteosynthesis presents a higher incidence of both intraoperative and postoperative complications compared to the implantation of primary total hip prostheses. Thus, while osteosynthesis remains a valuable intervention for femur fractures, careful attention to material selection and postoperative management is crucial in optimizing patient outcomes and minimizing complications.

DETAILED DESCRIPTION:
The aim was to identify the causes of mechanical failures of osteosynthesis in order to prevent them. Methods: We present the experience of the Department of Surgical Orthopedic Surgery, concerning 35 cases summarized after failure of surgical treatment of a fracture of the proximal end of the femur for a period spreading between January 2015 and December 2021. . The literature already found evidence of the greater complexity of this type of procedure compared to a first-line total hip prosthesis. Accordingly, all this, Prevention is better than cure these stiffnesses through good preoperative planning. Other factors related to the terrain or to untimely loading of the implant are more difficult to control. Whatever the cause, the surgeon remains by the rigor in these indications, the choice of the synthetic material the essential element in the prevention of osteosynthesis failures.

ELIGIBILITY:
Inclusion Criteria:

* • Diagnosis of a fracture of the proximal end of the femur.

  * Subsequent surgical intervention(s) due to failure of initial surgical treatment

Exclusion Criteria:

* • Those initially treated with total hip arthroplasty.

  * Patients lost to follow-up, not consistently monitored, or untreated after diagnosis of the complication.
  * Cases with incomplete medical records

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: cases of recurrent fractures of the proximal end of the femur following surgical treatment failure
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2021-12-02 (Actual)

PRIMARY OUTCOMES:
Surgical Approach | from enrollment to the of treatment 6 years
  type of approach
Preparation of the Patient | from enrollment to the of treatment 6 years
  type of preparation
Anesthesia | from enrollment to the of treatment 6 years
  type of anesthesia
Type of Surgical Revision | from enrollment to the of treatment 6 years
  material implanted for revision
Types of Prosthesis | from enrollment to the of treatment 6 years
  prothesis used

SECONDARY OUTCOMES:
Age Distribution | from enrollment to the end of treatment 6 years
  The average age of patients experiencing therapeutic failure after surgical treatment of proximal femur fractures was 66 years, with ages ranging from 28 to 94 years. The age group 50-90 years constituted 68.59% of cases.
Distribution by Sex | from enrollment to the end of treatment 6 years
  Females represented a slight majority in the study, accounting for 57% (20 women), while males comprised 43% (15 men).
Distribution According to Affected Side | from enrollment to the end of treatment 6 years
  The right side was affected in 60% (21 cases), while the left side was affected in 40% (14 cases).
Distribution According to Circumstances of Trauma | from enrollment to the end of treatment 6 years
  Fractures were predominantly due to minimal trauma, with rare occurrences related to road accidents or domestic falls, attributed to bone fragility and muscle atrophy. One case of a pathological fracture was observed in a patient with dislocation of an intermediate hip prosthesis due to ovarian cancer.

CONTACTS AND LOCATIONS:
Locations (1):
- IBN jazzar hospital, Kairouan, Tunisia

IPD SHARING:
Plan to Share IPD: No
use for other resaerchs